CLINICAL TRIAL: NCT07033702
Title: Pilot Study Assessing the Feasibility and Safety of the Airway Exchange Broncholaryngoscope (AEBLScope) During Routine Tracheostomy Tube Exchanges
Brief Title: Feasibility and Safety of the Airway Exchange Broncholaryngoscope (AEBLScope)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Karla O'Dell, Associate Professor of Otolaryngology - Head and Neck Surgery, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23-06016
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Tracheotomy Patients; Airway Management; Airway Disease
Keywords: tracheostomy; bronchoscope; airway exchange; feasibility; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Chronic Tracheostomy Tube-Dependent Patients (Experimental): All participants will be be chronically tracheostomy-tube dependent and undergo routine, in-office tracheostomy tube exchanges using the AEBLScope device.
  Interventions: Device: Airway-Exchange Broncholaryngoscope (AEBLScope)

INTERVENTIONS:
Device: Airway-Exchange Broncholaryngoscope (AEBLScope) — Airway Exchange Broncholaryngoscope (AEBLScope) - A modified disposable flexible bronchoscope designed to allow visualization during airway tube exchange procedures.

SUMMARY:
This pilot study evaluates the safety and feasibility of a novel airway exchange broncholaryngoscope (AEBLScope) during routine tracheostomy tube exchanges in chronically tracheostomy-dependent adult outpatients.

DETAILED DESCRIPTION:
The AEBLScope is a modified disposable bronchoscope designed to allow for simultaneous visualization during airway tube exchanges. This prospective, single-arm pilot study will assess the safety, feasibility, and effectiveness of the AEBLScope in low-risk airway tube exchanges.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Chronically (>1 month) tracheostomy-dependent outpatients
* Currently not requiring ventilatory or supplemental oxygen support
* Have undergone at least one prior tracheostomy tube exchange
* Scheduled for routine in-office tracheostomy tube exchange
* Able to provide informed consent

Exclusion Criteria:

* Active respiratory infection
* Patients with airway tubes having an inner diameter less than 6.0 mm
* Patients with preexisting pulmonary conditions, including chronic obstructive pulmonary disease (COPD), restrictive lung disease, untreated pneumonia, or acute respiratory distress syndrome (ARDS)
* Patients who are tracheostomy-dependent but cannot be orotracheally intubated.
* Patients unable to provide informed consent and who have no legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility - First-pass success rate of tracheostomy tube exchange using the AEBLScope | During procedure, at time of intervention
  First-pass success defined as successful tracheostomy tube placement on initial attempt using the AEBLScope without need for repeat attempt or alternative instrumentation.

SECONDARY OUTCOMES:
Feasibility - Procedure duration | During procedure, at time of intervention
  Duration of the airway exchange procedure using the AEBLScope measured in seconds from device insertion to device withdrawal.
Safety - Procedural complications | During procedure, at time of intervention
  Incidence of procedural complications related to use of the AEBLScope including but not limited to bleeding, airway trauma, patient intolerance, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Karla O'Dell, M.D., Principal Investigator — Univserity of Southern California
Locations (2):
- United States (2):
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roddy DJ, Spaeder MC, Pastor W, Stockwell DC, Klugman D. Unplanned Extubations in Children: Impact on Hospital Cost and Length of Stay. Pediatr Crit Care Med. 2015 Jul;16(6):572-5. doi: 10.1097/PCC.0000000000000406. PMID 25901542
- [Background] Needham DM, Pronovost PJ. The importance of understanding the costs of critical care and mechanical ventilation. Crit Care Med. 2005 Jun;33(6):1434-5. doi: 10.1097/01.ccm.0000166360.82336.75. No abstract available. PMID 15942375
- [Background] Tabaee A, Lando T, Rickert S, Stewart MG, Kuhel WI. Practice patterns, safety, and rationale for tracheostomy tube changes: a survey of otolaryngology training programs. Laryngoscope. 2007 Apr;117(4):573-6. doi: 10.1097/MLG.0b013e318030455a. PMID 17415123
- [Background] McLean S, Lanam CR, Benedict W, Kirkpatrick N, Kheterpal S, Ramachandran SK. Airway exchange failure and complications with the use of the Cook Airway Exchange Catheter(R): a single center cohort study of 1177 patients. Anesth Analg. 2013 Dec;117(6):1325-7. doi: 10.1213/ANE.0b013e3182a7cd3d. PMID 24257382
- [Background] Mort TC. Continuous airway access for the difficult extubation: the efficacy of the airway exchange catheter. Anesth Analg. 2007 Nov;105(5):1357-62, table of contents. doi: 10.1213/01.ane.0000282826.68646.a1. PMID 17959966
- [Background] Mort TC, Braffett BH. Conventional Versus Video Laryngoscopy for Tracheal Tube Exchange: Glottic Visualization, Success Rates, Complications, and Rescue Alternatives in the High-Risk Difficult Airway Patient. Anesth Analg. 2015 Aug;121(2):440-8. doi: 10.1213/ANE.0000000000000825. PMID 26111264
- [Background] Ng J, Hohman MH, Agarwal A. Tracheostomy Tube Change. 2024 Feb 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK555919/ PMID 32310379